CLINICAL TRIAL: NCT06908538
Title: Cryo NerVe Block Extremity AmputatioN RegIStry for Post Operative and pHantom Limb Pain (VANISH)
Brief Title: Cryo NerVe Block Extremity AmputatioN RegIStry for Post Operative and pHantom Limb Pain
Acronym: VANISH
Status: Recruiting | Type: Observational
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RP-2025-0001
Record Dates: First submitted 2025-03-19; First posted 2025-04-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-03

CONDITIONS: Amputation; Amputation of Lower Limb; Amputation of Upper Limb; Amputation, Limb Loss; Amputation, Traumatic/Surgery; Cryo Analgesia
MeSH Terms: interventions — Cryosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects who have or will have an amputation procedure.: The primary objective of this Registry is to capture real-world safety and performance data on AtriCure devices used to cryoablate nerves during an extremity amputation procedure.
  Interventions: Device: cryoablation

INTERVENTIONS:
Device: cryoablation — Cryoanalgesia, also known as Cryoablation, Cryoneurolysis, or Cryonerve Block, has been used for decades to treat chronic pain and has recently been employed for the management of Phantom Limb Pain. Cryoanalgesia involves the use of a probe to apply extreme cold (approximately -70◦C) to induce reversible axonal injury and Wallerian degeneration to produce a temporary conduction block that is sustained until regeneration of the axon and sensation is restored, typically weeks to months later.

SUMMARY:
The goal of this Registry is to see how the device is used when freezing nerves during an amputation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have or will have an amputation procedure;
* Patients who are willing and capable of providing informed consent;
* Patients whose age is 18 years or above, or of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

* Women of childbearing potential who are, or plan to become, pregnant during the time of the study;
* Other medical, social, or psychological conditions that in the opinion of the Investigator precludes the subject from appropriate consent or adherence to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have or will have an amputation procedure.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2035-04 (Estimated); Study Completion 2035-04 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 30 days
  CryoNerve Block procedural complications

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Elliot Hospital, Manchester, New Hampshire
  - NYU Langone Health, New York, New York
  - Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided